CLINICAL TRIAL: NCT00004224
Title: SIOP Study of Combined Modality Treatment in Childhood Ependymoma
Brief Title: Combination Chemotherapy Followed by Radiation Therapy in Treating Children With Localized Ependymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Societe Internationale d'Oncologie Pediatrique (Other)
Collaborators: Children's Cancer and Leukaemia Group (Other); Italian Association for Pediatric Hematology Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067465; SIOP-EPENDYMOMA-99; AIEOP-EPENDYMOMA-99; CCLG-EPENDYMOMA-99; EU-99001
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood infratentorial ependymoma; childhood supratentorial ependymoma; newly diagnosed childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Cyclophosphamide; Etoposide; Vincristine; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: etoposide
Drug: vincristine sulfate
Procedure: adjuvant therapy
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug and combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying combination chemotherapy and radiation therapy to see how well they work in treating children with localized ependymoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the event free and overall survival of children with incompletely resected localized ependymoma when treated with adjuvant cyclophosphamide, etoposide, and vincristine followed by radiotherapy.
* Determine the response rate in these patients to this regimen.

OUTLINE: This is a multicenter study.

Patients undergo surgery to remove as much of tumor as possible. Patients with residual disease proceed to chemotherapy, while those with no residual disease proceed directly to radiotherapy.

Chemotherapy begins within 3 weeks of surgery and consists of vincristine IV on days 1, 8, and 15, cyclophosphamide IV over 3 hours on day 1, and etoposide IV over 4 hours on days 1-3. Treatment repeats every 4 weeks for up to 4 courses. Patients who progress after 2 courses proceed to radiotherapy. If residual disease is still present at completion of chemotherapy, second look surgery is recommended.

Patients undergo radiotherapy daily for 6 weeks beginning after complete resection within 4 weeks of surgery, within 3 weeks of completion of chemotherapy, or within 4 weeks of second look surgery.

Patients are followed at 6 weeks after radiotherapy, every 2 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven nonmetastatic intracranial ependymoma

  * Cellular
  * Papillary
  * Clear cell
  * Mixed cell
  * Anaplastic
* No myxopapillary ependymoma, subependymoma, or ependymoblastoma

PATIENT CHARACTERISTICS:

Age:

* 3 to 20

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* No hematologic disease that would preclude study participation

Hepatic:

* Not specified

Renal:

* No renal disease that would preclude study participation

Other:

* No concurrent unrelated disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior steroids allowed

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 1999-01; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Event-free survival
Overall survival
Surgical operability
Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Richard Grundy, MD, PhD, Study Chair — Birmingham Children's Hospital; Maura Massimino, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (7):
- Fundacion para la Lucha contra las Enfermedades Neurologicas de la Infancia, Buenos Aires, Buenos Aires, Argentina
- Hospital for Sick Children, Toronto, Ontario, Canada
- Fondazione Istituto Nazionale dei Tumori, Milan, Italy
- Erasmus MC - Sophia Children's Hospital, Rotterdam, Netherlands
- Hospital Des Cruces, Vizcaya, Spain
- Ostra Sjukhuset, Gothenburg, Sweden
- Birmingham Children's Hospital, Birmingham, England, United Kingdom